CLINICAL TRIAL: NCT06949514
Title: The Effect of Guided Imagery on Anxiety, Depression, and Sleep in Hospitalized Pregnant Women
Brief Title: Guided Imagery in Hospitalized Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menekşe Nazlı AKER (Other)
Responsible Party: Sponsor-Investigator, Menekşe Nazlı AKER, Assist. Prof., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 06.01.2025/01-14
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Guided imagery group
  Interventions: Other: guided imagery
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Other: guided imagery — Participants in this group will receive the guided imagery intervention. They will be approached after being hospitalized for at least 24 hours. The guided imagery audio recording will be played for the pregnant women every evening before sleep for three consecutive days.
  Arms: Intervention Group

SUMMARY:
The study will be carried out in two different groups. Participants will be approached after being hospitalized for at least 24 hours. After the pregnant women are evaluated in terms of eligibility criteria for the research, the pregnant women who are eligible will be informed about the research and written informed consent will be obtained from the pregnant women who accept. The random distribution of pregnant women to the study groups will be carried out random.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having no difficulties in understanding and speaking Turkish
* Being hospitalized for at least 24 hours
* Being in the second trimester of pregnancy (14-28 weeks)
* Having a medically stable condition
* Experiencing sleep disturbances
* Voluntarily agreeing to take part in the study

Exclusion Criteria:

* Having a hearing impairment
* Having ongoing severe vaginal bleeding
* Having a diagnosed psychiatric disorder and/or using psychiatric medication
* Having uncontrolled hypertension
* Presence of intrauterine fetal demise
* Premature rupture of membranes (PROM)
* Being in preterm labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | at the beginning of the study, 3 days later
  The Hospital Anxiety and Depression Scale is a four-point Likert-type scale used to determine the risk, level, and change in severity of anxiety and depression in patients. The scale consists of 14 items; odd-numbered items assess anxiety, and even-numbered items assess depression. For the anxiety subscale, the cut-off score is 10/11. Individuals scoring above this threshold are considered to be at risk. The lowest possible score on the scale is 0, and the highest possible score is 21.
Change in Depression | at the beginning of the study, 3 days later
  The Hospital Anxiety and Depression Scale is a four-point Likert-type scale used to determine the risk, level, and change in severity of anxiety and depression in patients. The scale consists of 14 items; odd-numbered items assess anxiety, and even-numbered items assess depression. For the depression subscale, the cut-off score is 7/8. Individuals scoring above this threshold are considered to be at risk. The lowest possible score on the scale is 0, and the highest possible score is 21.
Change in Sleep Quality | at the beginning of the study, 3 days later
  The Richard-Campbell Sleep Questionnaire consists of six items that evaluate the depth of night sleep, time taken to fall asleep, frequency of awakenings, duration of wakefulness upon awakening, overall sleep quality, and the level of noise in the environment. Each item is assessed using a visual analog scale ranging from 0 to 100. Scores between 0-25 indicate very poor sleep, while scores between 76-100 indicate very good sleep. As the total score increases, the sleep quality of patients also improves.

CONTACTS AND LOCATIONS:
Overall Officials: Menekşe Nazlı Aker, Study Director — Assistant professor
Locations (1):
- Aksaray Eğitim Araştırma Hastanesi, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No